CLINICAL TRIAL: NCT05243173
Title: Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Brief Title: Biomarkers of Response to Systemic Treatments in FH-deficient RCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RJFHRCC
Record Dates: First submitted 2021-12-20; First posted 2022-02-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Metabolomics; Renal Cell Carcinoma; FH-Deficient RCC; Systemic Treatments
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tumor tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sequencing — Laboratory analysis of samples

SUMMARY:
Fumarate hydratase-deficient renal cell carcinoma (FH-deficient RCC) is a rare subtype of RCC characterized by germline/somatic mutation of the fumarate hydratase (FH) gene, and is an extremely aggressive tumor, with a propensity to disseminate early even in the setting of a small primary tumor.

Affected individuals or individuals suspected of having a germline FH will undergo periodic clinical assessment and genetic analyses for the purpose of: 1) definition and characterization of phenotype, 2) determination of the natural history of the disorder, and 3) genotype/phenotype correlation. Genetic linkage studies may be performed in situations in which the genetic basis of the disorder has not been elucidated.

DETAILED DESCRIPTION:
* Discovery and validation of biomarker predicting FH-deficient RCC systemic treatments response
* Analysis for expression level of ctDNA using Next generation sequencing in FH-deficient RCC blood by systemic treatments response
* Analysis for expression level of mRNA using Next generation sequencing in FH-deficient RCC tissue by systemic treatments response
* Analysis for expression level of small molecule metabolites using mass spectrometry in FH-deficient RCC tissue and blood by systemic treatments response
* Analysis for genetic and protein expression at a single-cell level using a novel flow cytometry and RNA-sequencing protocol in FH-deficient RCC tissue and blood.
* Validation of genetic and protein expression using qRT-PCR or IHC in multiple independent cohort.
* Biological biomarkers-clinical factor combined prediction model of FH-deficient RCC systemic treatments response

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. histopathological evidence of FH-deficient renal cell carcinoma, which was confirmed by Sanger or next-generation sequencing after initial screening by IHC.
3. included patients must be diagnosed with metastatic renal cell carcinoma or have a TNM stage IV (according to 2009 TNM Classification);
4. new FH-RCC patients who has scheduled to start 1st cycle of systemic treatment;
5. ECOG score ≤2;
6. life expectancy ≥ 3 months;
7. sign informed consent, and be able to follow the visit and related procedures stipulated in the program;
8. agree to collect tumor tissue, blood and other specimens required by this study and apply them to relevant studies;
9. Patients must have consent in place, for the use of tissue and imaging to be used for the purposes of clinical research; Use of tissue not required for their diagnosis or treatment to be stored and used for the purposes of clinical research, which may include genetic research. Use of relevant sections of their medical records, or by relevant regulatory authorities, where my tissue is being used for research, giving permission for those individuals to have access to their medical records. Participants must also meet at least one of the following criteria to be eligible: For tissue analysis: Patient must have tumour tissue and/or normal adjacent kidney stored (either as formalinfixed paraffin-embedded tissue, or as 'fresh frozen' tissue). For imaging analysis: Patient must have had at least 1 scan (either CT or MRI) within 28 days of starting treatment with systemic treatment for their cancer.

Exclusion Criteria:

1. patients with other malignant tumors with different primary sites or histology from the tumor evaluated in this study within 2 years of personal history, except those with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or cervical carcinoma in situ under good control;
2. major surgery or severe trauma within 4 weeks before enrollment;
3. known or suspected active autoimmune diseases (congenital or acquired), such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. Patients with type 1 diabetes with good insulin control can also be enrolled.
4. known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
5. allergic to any component of monoclonal antibody;
6. suffering from other uncontrolled serious diseases, including but not limited to: A) severe infection in the active phase or clinically poorly controlled; B) HIV infection (HIV antibody positive); C) acute or chronic active hepatitis b (HBsAg positive and HBV DNA>1*103/ml) or acute or chronic active hepatitis c (HCV antibody positive and HCV RNA>15IU/ml); D) active tuberculosis, etc.;
7. class iii-iv congestive heart failure (New York heart association classification), poorly controlled and clinically significant arrhythmia;
8. uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg);
9. pregnant or lactating women.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with FH-RCC who have given prior consent for their samples and data to be used, and who have adequate samples and data available.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | 2 years
  across multiple LC-MS data files. across multiple LC-MS data files. across multiple LC-MS data files. across multiple LC-MS data files. across multiple LC-MS data files
Determine genotype/phenotype correlations | 3 years
  Collection of blood, tissue & urine to address further scientific questions related to this protocol.
Discovery of predicting bio-markers for FH-deficient RCC systemic treatments response | 3 years
  Combination prediction model of biologic biomarkers and clinical factors for the response of systemic treatments in FH-RCC.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunze Xu, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided